CLINICAL TRIAL: NCT01903369
Title: Comparison of Intraneural and Extraneural Young's Modulus Using Shear Wave Elastography in Patients Undergoing Regional Anaesthesia
Brief Title: Comparison of Intraneural and Extraneural Young's Modulus Using Shear Wave Elastography
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: Tenovus 13/7
Record Dates: First submitted 2013-07-11; First posted 2013-07-19 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Regional Anaesthesia
Keywords: Shear wave; Elastography; Repeatability and Reproducibility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Elective orthopaedic surgery patients: All patients presenting for elective orthopaedic surgery >16 years of age.
  Interventions: Device: Shear Wave Elastography

INTERVENTIONS:
Device: Shear Wave Elastography — Shear wave elastography
  Other Names: Siemens 3000 shear wave utrasound machine

SUMMARY:
The investigators would like to compare the stiffness inside and outside nerves using a special type of ultrasound imaging called shear wave elastography. Shear wave elastography is a special form of ultrasound as the pictures taken are in colour. An ultrasound machine has different ways of taking pictures of inside the body: one is by measuring the brightness of different body parts (often referred to as the B-Mode scan), the pictures taken in this way are the same as those you may have seen of unborn babies inside their mum's tummies; another way is by measuring the stiffness of different body structures which is how shear wave elastography works. The investigators hope that this new technology will help doctors to see the parts of the body that are important to them.

DETAILED DESCRIPTION:
Shear wave elastography is a quantitative ultrasound modality increasingly used to differentiate between "hard" breast cancer masses and "soft" normal tissue. Unlike strain elastography, shear wave elastography applies a non-compressive longitudinal acoustic radiation force to underlying tissues, inducing transverse shear waves. Studies in Thiel embalmed human cadavers have shown significant differences in Young's modulus between intraneural and extraneural tissue, and ready colour differentiation between tissues.

The investigators own pilot studies have shown a 3-fold greater Young's modulus within nerve in Thiel embalmed cadavers and human volunteers. The investigators hypothesis is that shear wave elastography can differentiate between nerve and adjacent tissue in patients before nerve block for surgery. If so, this technology has the potential to reduce the incidence of complications with UGRA and encourage parallel applications such as cancer node biopsy.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for elective orthopaedic surgery >16 years of age.
* ASA score 1, 2 or 3.
* Capacity to provide informed consent.

Exclusion Criteria:

* Patients not undergoing ultrasound guided regional anaesthesia.
* ASA score 4 or above.
* Patients without the capacity to provide informed consent.
* Pregnant women.
* Patients currently participating in another research project or patients who have participated in a research project in the 6 months

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing routine ultrasound-guided regional anaesthesia for elective orthopaedic surgery at Ninewells Hospital & Medical School, Dundee.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2015-03-26 (Actual); Study Completion 2015-07-10 (Actual)

PRIMARY OUTCOMES:
The difference in stiffness between nerves and surrounding tissue in patients when using shear wave measurement before regional anaesthesia. | One visit per patient 45 mins
  Youngs modulus

CONTACTS AND LOCATIONS:
Overall Officials: Graeme A McLeod, MBChB FRCA, Principal Investigator — NHS Tayside
Locations (1):
- Department of Anaesthesia, Ninewells Hospital & Medical School, Dundee, United Kingdom

REFERENCES:
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Background] Neal JM, Brull R, Chan VW, Grant SA, Horn JL, Liu SS, McCartney CJ, Narouze SN, Perlas A, Salinas FV, Sites BD, Tsui BC. The ASRA evidence-based medicine assessment of ultrasound-guided regional anesthesia and pain medicine: Executive summary. Reg Anesth Pain Med. 2010 Mar-Apr;35(2 Suppl):S1-9. doi: 10.1097/AAP.0b013e3181d22fe0. PMID 20216019
- [Background] Neal JM, Wedel DJ. Ultrasound guidance and peripheral nerve injury: is our vision as sharp as we think it is? Reg Anesth Pain Med. 2010 Jul-Aug;35(4):335-7. doi: 10.1097/AAP.0b013e3181e8a3bb. No abstract available. PMID 20588150
- [Background] Liu SS, YaDeau JT, Shaw PM, Wilfred S, Shetty T, Gordon M. Incidence of unintentional intraneural injection and postoperative neurological complications with ultrasound-guided interscalene and supraclavicular nerve blocks. Anaesthesia. 2011 Mar;66(3):168-74. doi: 10.1111/j.1365-2044.2011.06619.x. PMID 21320084
- [Background] Palmeri ML, Dahl JJ, MacLeod DB, Grant SA, Nightingale KR. On the feasibility of imaging peripheral nerves using acoustic radiation force impulse imaging. Ultrason Imaging. 2009 Jul;31(3):172-82. doi: 10.1177/016173460903100303. PMID 19771960
- [Background] Wells PN, Liang HD. Medical ultrasound: imaging of soft tissue strain and elasticity. J R Soc Interface. 2011 Nov 7;8(64):1521-49. doi: 10.1098/rsif.2011.0054. Epub 2011 Jun 16. PMID 21680780
- [Background] Evans A, Whelehan P, Thomson K, McLean D, Brauer K, Purdie C, Jordan L, Baker L, Thompson A. Quantitative shear wave ultrasound elastography: initial experience in solid breast masses. Breast Cancer Res. 2010;12(6):R104. doi: 10.1186/bcr2787. Epub 2010 Dec 1. PMID 21122101
- [Background] Munirama S, Joy J, Eisma R, Corner G, Cochran S, McLeod G. Shear wave elastography: novel technology for ultrasound-guided regional anesthesia. Anesthesiology. 2013 Sep;119(3):698. doi: 10.1097/ALN.0b013e31827ddeb6. No abstract available. PMID 23291624
- [Background] Arda K, Ciledag N, Aktas E, Aribas BK, Kose K. Quantitative assessment of normal soft-tissue elasticity using shear-wave ultrasound elastography. AJR Am J Roentgenol. 2011 Sep;197(3):532-6. doi: 10.2214/AJR.10.5449. PMID 21862792